CLINICAL TRIAL: NCT02902588
Title: The Use of Near Infrared Spectroscopy and Magnetic Resonance Imaging Technique in the Evaluation of the Permeability of Blood-brain Barrier in Adults With Meningitis
Brief Title: Blood-brain Barrier Permeability Study in Adults With Meningitis
Acronym: NM-BBBP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The tests have been completed
Sponsor: Nalecz Institute of Biocybernetics and Biomedical Engineering, Polish Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: BBBP-1PW5
Record Dates: First submitted 2016-08-23; First posted 2016-09-16 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Blood-Brain Barrier Permeability
Keywords: Blood-Brain Barrier; Magnetic Resonance Imaging; Spectroscopy, Near-Infrared; Indocyanine green
MeSH Terms: interventions — Gadolinium; gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ICG washout kinetics assessment (Experimental): Intravenous administration of 5-10 mg indocyanine green (ICG-PULSION), once per subject
  Interventions: Other: ICG-PULSION
- Pulse oximeter monitor (Other): Monitoring of a person's oxygen saturation (SO2), peripheral oxygen saturation
  Interventions: Device: LiMON, Pulsion Medical Systems
- Gadolinium washout kinetics assessment (Experimental): 20 mL of gadolinium (Gadovist, Bayer, Germany) injection at 5 mL/s, once per subject
  Interventions: Other: Gadolinium (Gadovist, Bayer, Germany)

INTERVENTIONS:
Other: ICG-PULSION — Intravenous administration of indocyanine green
  Arms: ICG washout kinetics assessment
Device: LiMON, Pulsion Medical Systems — Application of near infrared light
  Arms: Pulse oximeter monitor
Other: Gadolinium (Gadovist, Bayer, Germany) — Injection of gadolinium
  Arms: Gadolinium washout kinetics assessment

SUMMARY:
The purpose of the study is to confirm the applicability and usefulness of the novel method of assessment of the permeability of the blood-brain barrier and in monitoring of the treatment of patients with meningitis. The proposed technique is based on evaluation of the kinetics of the indocyanine green (ICG) outflow from the brain with the use of near-infrared spectroscopy (NIRS). Usefulness of the NIRS-based method will be analyzed in relation to the reference method, which is contrast-enhanced magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Clinical trials in healthy volunteers and in patients with diagnosed blood-brain barrier disruption:

* Performing a lumbar puncture as a routine diagnostic procedure in a patient with suspected neuroinfection. Biochemical assessment of the degree of the blood-brain barrier disruption based on the albumin ratio.
* Enrollment of patients diagnosed with neuroinfection to the study and obtaining informed consent.
* Performing the measurement involving fixation of the NIRS probes on the patient's head while intravenously injecting optical contrast agent - ICG (5-10 mg in a bolus). The measurement time is about 15 min. Monitoring of the patient's condition during the examination using a pulse oximeter monitor. The examination should be performed no later than 12 hours after the lumbar puncture to obtain a reliable correlation of results between the methods. The party responsible for the technical aspect of the investigation will be the Sponsor while the party responsible for the medical aspect (including the injection of the contrast agent) will be the Principal Investigator.
* Conducting a magnetic resonance test. The MRI imaging can be carried out before or after the test by the optical method, but with only a slight time delay (not more than 24h). The gadolinium will be injected at 5 mL/s (20 mL per patient). Calculating the cerebral blood flow and the cerebrovascular permeability coefficient and passing the information to the patient's doctor.

  3. The assessment of the contrast agent outflow kinetics parameters obtained with use of the optical method 4. The correlation of the results of the of the evaluation of the blood-brain barrier condition by MRI, biochemical assessment of the cerebro-spinal fluid and optical method.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* diagnosed with meningitis in the examination of cerebrospinal fluid

Exclusion Criteria:

* allergic to any of the contrast agents
* a lack of consent to the test
* liver failure and kidney failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Correlation between blood brain barrier permeability assessment with use of near infrared spectroscopy and magnetic resonance imaging | up to 12 months
  The kinetics of the indocyanine green (ICG) outflow from the brain with the use of near-infrared spectroscopy will be a subject of investigation. ICG washout rate parameter R [a.u.] will be calculated which describes the effectiveness of the washout of ICG from the brain. It is calculated by measuring the accumulation of ICG contrast agent in the extravascular-extracellular space. The volume transfer constant (Ktrans) which reflects the efflux rate of gadolinium contrast from blood plasma into the tissue extravascular-extracellular space will be assessed during contrast-enhanced magnetic resonance imaging study. Ktrans is a measure of capillary permeability. Both parameters may reflect blood brain barrier (BBB) permeability and indicate BBB disruption. The primary outcome of the study will be correlation coefficient r [a.u.] between R and Ktrans calculated for the set of subjects. Adverse events as a consequence of ICG and/or gadolinium administration will be monitored and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Liebert, Prof., Study Chair — Nalecz Institute of Biocybernetics and Biomedical Engineering Polish Academy of Science
Locations (1):
- Medical University in Bialystok, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ergin A, Wang M, Zhang JY, Bruce JN, Fine RL, Bigio IJ, Joshi S. The feasibility of real-time in vivo optical detection of blood-brain barrier disruption with indocyanine green. J Neurooncol. 2012 Feb;106(3):551-60. doi: 10.1007/s11060-011-0711-5. Epub 2011 Oct 1. PMID 21964696
- [Result] Liebert A, Milej D, Weigl W, Gerega A, Kacprzak M, Maniewski R. Fluorescence-based method for assessment of blood-brain barrier disruption. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:3040-2. doi: 10.1109/EMBC.2013.6610181. PMID 24110368